CLINICAL TRIAL: NCT04740892
Title: A Clinical Evaluation of the Safety and Efficacy of a Moisturizing Cream and Baby Wash in the Management of Mild to Moderate Atopic Dermatitis in Infants, Toddlers and Children
Brief Title: A Study of a Moisturizing Cream and Baby Wash in the Management of Mild to Moderate Atopic Dermatitis in Infants, Toddlers and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSSKB003103; CCSSKB003103 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-01-21; First posted 2021-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wash and Cream Investigational Product (IP) (Experimental): Parent participant will bathe the child participant with the investigational wash at least 3 times per week, but no more than once daily, for 4 weeks. Parent participant will apply the investigational cream on their child participant twice daily for 4 weeks.
  Interventions: Other: Wash IP; Other: Cream IP

INTERVENTIONS:
Other: Wash IP — Parent participant will bathe the child participant with the investigational wash at least 3 times per week, but no more than once daily, for 4 weeks.
Other: Cream IP — Parent participant will apply the investigational cream on their child participant twice daily for 4 weeks.

SUMMARY:
The purpose of this study is to evaluate the effectiveness (assessed by clinical evaluation of eczema/atopic dermatitis severity and parent-perceived benefits) and tolerability (assessed by clinical grading and parent-perception) of the investigational cream when used in conjunction with a baby wash in babies, toddlers, and children with mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

For Child

* Fitzpatrick skin type I to VI
* Child must have at least 1 target lesion based on the atopic dermatitis severity index (ADSI) with a score of 2-12 and an erythema sub score of at least 2 (moderate)
* Has mild to moderate atopic dermatitis (as per Rajka-Langeland Severity Index; graded as 3.0 to 7.5 inclusive)
* Child must have parent-assessed history of itch
* Has parent-perceived sensitive skin For Parents
* Willing to undergo a 3-day washout period prior to the baseline assessments. During this run-in period, parents will be asked to refrain from using prescription and over-the-counter (OTC) eczema treatments on their child; Acute rescue treatment will be permitted (type of rescue treatment will be determined by principal investigator [PI])
* Has signed the informed consent document (ICD), including Health Insurance Portability and Accountability Act (HIPAA) disclosure

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products or ingredients of the investigational products (IPs)
* Has a history of a confirmed or suspected coronavirus disease 2019 (COVID-19) infection within 30 days prior to Visit 1 For Child
* Presents with a skin condition that may influence the outcome of the study (specifically psoriasis or active skin cancer)
* Severe atopic dermatitis (AD) as determined by the Rajka-Langeland Severity Index For Parent
* Is self-reported to be pregnant or planning to become pregnant during the study

Ages: 3 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Eczema Area Severity Index (EASI) After 4 Weeks of Product Use | Baseline, Week 4
  EASI is a composite scoring system index which is used to measure the severity of 4 clinical manifestations of atopic dermatitis (erythema, edema/induration/papulation, excoriations, and lichenification) according to the percentage of affected area in each of the 4 body regions (head/neck, trunk, upper limbs, and lower limbs). Final scores range from 0 (no disease anywhere on the body) to 72 (severest disease on all body areas).
Change From Baseline in Atopic Dermatitis Severity Index (ADSI) After 4 Weeks of Product Use | Baseline, Week 4
  ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a scale of 0 (none) to 3 (severe). The total score can range from 0 (no eczema signs) to 15 (severe eczema lesion).

SECONDARY OUTCOMES:
Change From Baseline in Skin Microbiome | Baseline, Day 1, 3, 7 and Week 4
  Change from baseline in skin microbiome in lesion versus adjacent non-lesional site will be assessed. Microbiome samples collected from the identified lesional site and an adjacent non-lesional site by swabbing technique will be analyzed by using 16s ribonucleic acid (RNA) sequencing.
Change From Baseline in EASI | Baseline, Day 1, 3 and 7
  EASI is a composite scoring system index which is used to measure the severity of 4 clinical manifestations of atopic dermatitis (erythema, edema/induration/papulation, excoriations, and lichenification) according to the percentage of affected area in each of the 4 body regions (head/neck, trunk, upper limbs, and lower limbs). Final scores range from 0 (no disease anywhere on the body) to 72 (severest disease on all body areas).
Change From Baseline in ADSI | Baseline, Day 1, 3 and 7
  ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a scale of 0 (none) to 3 (severe). The total score can range from 0 (no eczema signs) to 15 (severe eczema lesion).
Change From Baseline in Caregiver Itch Assessment Score | Baseline, Day 1, 3, 7 and Week 4
  Parent participant will assess how much itching/scratching the child participant has been exhibiting on a scale of 1 (none) to 4 (all the time). An option of "I don't have an opinion" will be included.
Change From Baseline in Infant Dermatitis Quality of Life Index (IDQoL) | Baseline, Day 1, 3, 7 and Week 4
  IDQoL is a validated questionnaire completed by parents to assess the impact of atopic dermatitis on the quality of life in infants aged 0-3 years. The Infant's Dermatitis Quality of Life Index is calculated by summing the score of each question: for question 1 (0 [none] to 3 [all the time]), For question 2 (0 [happy] to 3 [always crying]), For question 3 (0 [0-15 minutes to 3 [More than 2 hours]), For question 4 (0 [less than one hour] to 3 [Five hours or more]), and For questions 5 to 10 (0 [None] to 3 [Very much]), resulting in a maximum score of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The severity of eczema is scored separately and can be correlated with the Infants' Dermatitis Quality of Life Index. The score of Dermatitis severity ranges from 0 (None) to 4 (Extremely severe).
Change From Baseline in Brief Infant Sleep Questionnaire-Revised (BISQ-R) Scale Score | Baseline, Day 1, 3, 7 and Week 4
  BISQ-R is an age-based, norm-referenced scoring system that provides a comprehensive assessment of infant and toddler sleep patterns. Five (5) items related to sleep onset latency, number, and duration of night wakings, longest stretch of sleep and total night sleep. Parent perception consists of 3 items related to bedtime difficulty, overnight sleep, and overall child sleep problems. Parent behaviors consisting of 11 items related to bedtime routine consistency, bedtime, parental behavior at time of sleep onset and night wakings, sleep locations at time of sleep onset and following night wakings that may impact sleep outcomes. Score ranging from 0-100 is derived for each sub-scale, with higher scores denoting better sleep quality, more positive perceptions of sleep quality, and parental habits that promote healthy sleep behaviors and independent infant sleep, respectively. Total score is calculated as an average of infant sleep, parent perceptions and parent behavior subscale scores.
Parent Perceived Product Efficacy as Assessed by Parental Questionnaire | Baseline (immediately after first use) and Week 4
  Parent perceived product efficacy will be assessed by using parental questionnaire. Participant responses for each question will have 5 response options, the following numerical assignment could be one of the following choices: (1) Strongly Disagree, (2) Disagree Somewhat, (3) Neither Disagree or Agree, (4) Agree Somewhat, (5) Strongly Agree.
Change From Baseline in Transepidermal Water Loss (TEWL) Measurement in Lesion and Adjacent Non-lesional Site | Baseline, Day 1, 3, 7 and Week 4
  Change from Baseline in TEWL measurement on both the identified lesional site and an adjacent or non-lesional site will be reported. The DermaLab TEWL instrument uses a non-invasive probe, which measures the passive transfer of water through the stratum corneum.
TEWL Measurement Difference Between Lesion and Adjacent Non-lesional Site | Day 1, 3, 7 and Week 4
  TEWL measurement difference between lesional site and an adjacent non-lesional site will be reported. The DermaLab TEWL instrument uses a non-invasive probe, which measures the passive transfer of water through the stratum corneum.
Change from Baseline in Skin Hydration in Lesion and Adjacent Non-lesional Site | Baseline, Day 1, 3, 7 and Week 4
  Change from Baseline in skin hydration on both the identified lesional site and an adjacent or non-lesional site will be reported. The DermaLab hydration instrument uses a non-invasive probe, which measures the water content of the stratum corneum.
Skin Hydration Difference between Lesion and Adjacent Non-lesional Site | Day 1, 3, 7 and Week 4
  Skin hydration difference between lesion and adjacent non-lesional site will be reported. The DermaLab hydration instrument uses a non-invasive probe, which measures the water content of the stratum corneum.
Change From Baseline in Skin pH in Lesion Versus Adjacent Non-lesional Site | Baseline, Day 1, 3, 7 and Week 4
  Change from Baseline in skin pH on both the identified lesional site and an adjacent or non-lesional site will be reported. The DermaLab skin pH instrument uses a non-invasive probe, which measures the pH of the stratum corneum.
Skin pH Difference between Lesion and Adjacent Non-lesional Site | Day 1, 3, 7 and Week 4
  Skin pH difference between lesion and adjacent non-lesional site will be reported. The DermaLab skin pH instrument uses a non-invasive probe, which measures the pH of the stratum corneum.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Diana Draelos, MD, Principal Investigator — Dermatology Consulting Services, PLLC; Laura M Brooks, M.D., Principal Investigator — The Education & Research Foundation, Inc.
Locations (2):
- United States (2):
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Lipozencic J, Wolf R. Atopic dermatitis: an update and review of the literature. Dermatol Clin. 2007 Oct;25(4):605-12, x. doi: 10.1016/j.det.2007.06.009. PMID 17903619
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Rajka G, Langeland T. Grading of the severity of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1989;144:13-4. doi: 10.2340/000155551441314. PMID 2800895
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Basra MK, Gada V, Ungaro S, Finlay AY, Salek SM. Infants' Dermatitis Quality of Life Index: a decade of experience of validation and clinical application. Br J Dermatol. 2013 Oct;169(4):760-8. doi: 10.1111/bjd.12563. PMID 23909890
- [Background] National Psoriasis Foundation, "Topical Steriods Potency Chart," 18 December 2020, [Online]. Available: http;//www.psoriasis.org/potency_chart/.
- [Background] Avi Sadeh, D. Sc., Jodi A. Mindell, Ph.D., and Liat Tikotzky, Ph.D. Brief Infant Sleep Questionnaire - Revised Long Form, version January 2020
- See also: A Clinical Evaluation of the Safety and Efficacy of a Moisturizing Cream and Baby Wash in the Management of Mild to Moderate Atopic Dermatitis in Infants, Toddlers and Children — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKB003103&attachmentIdentifier=9c9d8dd0-9db7-4a25-acf0-86f4e38cc6f5&fileName=CCSSKB003103_CSR_Synopsis_English.pdf&versionIdentifier=